CLINICAL TRIAL: NCT03719820
Title: Stroke Imaging Package Study of Intracranial Atherosclerosis
Brief Title: Stroke Imaging Package Study of Intracranial Atherosclerosis ( SIPS-ICAS )
Acronym: SIPS-ICAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wei-Hai Xu (Other)
Collaborators: Peking Union Medical College Hospital (Other); General Hospital of Chinese Armed Police Forces (Other); General Hospital of Shenyang Military Region (Other); Subei People's Hospital of Jiangsu Province (Other); Fujian Medical University Union Hospital (Other); Tangshan Gongren Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Qingdao Municipal Hospital (Other); West China Hospital (Other); Shanghai Tong Ren Hospital (Other); Ruijin Hospital (Other); The First Affiliated Hospital of University of South China (Other); JiNing NO.1 People Hospital (Unknown); Tongji Hospital (Other); The University of HongKong-Shenzhen Hospital (Unknown); Beijing Anzhen Hospital (Other); Beijing Hospital (Other Government); Peking University International Hospital (Other); Beijing Tongren Hospital (Other); China-Japan Friendship Hospital (Other); Peking University First Hospital (Other); Beijing Friendship Hospital (Other); Beijing Chao Yang Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other); Shandong Provincial Hospital (Other Government); The Second Hospital of Hebei Medical University (Other); Hebei General Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); China-Japan Union Hospital, Jilin University (Other); Zhejiang Provincial Tongde Hospital (Other); People's Hospital of Ningxia Hui Autonomous Region (Other); Taiyuan Central Hospital of Shanxi Medical University (Other); Hong Xinglong Central Hospital (Unknown); Changzhi People's Hospital (Other); Weihai Municipal Hospital (Other); Southwest Hospital, China (Other); Affiliated Taihe Hospital of Hubei University of Medicine (Unknown); Nanshi Hospital of Nanyang (Unknown)
Responsible Party: Sponsor-Investigator, Wei-Hai Xu, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: HRMRI II
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Acute Ischemic Stroke AIS; Intracranial Atherosclerosis ICAS
Keywords: Acute Ischemic Stroke; Intracranial Atherosclerosis ICAS; HRMRI
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin; Clopidogrel; Rosuvastatin Calcium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intracranial Atherosclerosis: First-ever stroke patients attributed to intracranial artery stenosis (> 50% or occlusion) who receive aggressive medical management
  Interventions: Drug: aggressive medical management

INTERVENTIONS:
Drug: aggressive medical management — Aspirin (100 mg daily) and Clopidogrel (75 mg daily) for 3 months and Rosuvastatin (20mg daily) for at least 6 months as well as traditional risk factors management
  Other Names: Aspirin; Clopidogrel; Rosuvastatin

SUMMARY:
A prospective, multicenter, cohort study to explore the stroke mechanisms of symptomatic intracranial atherosclerosis, the dynamic changes under aggressive medical treatment and their associations with clinical events using conventional MRI sequences plus high-resolution magnetic resonance (HR-MRI).

DETAILED DESCRIPTION:
1. First-ever stroke patients attributed to intracranial artery stenosis (> 50% or occlusion) within 7 days after onset will be prospectively enrolled in our study and undergo new imaging technique package assessment at baseline.
2. The imaging technique package includes conventional cranial MRI （T1,T2,T2 FLAIR,DWI), cranial magnetic resonance angiography (MRA),high-resolution magnetic resonance (HR-MRI) and susceptibility weighted imaging (SWI) or T2*-weighted imaging.
3. Enrolled patients are recommended to receive aggressive medical management consisted of Aspirin (100 mg daily) and Clopidogrel (75 mg daily) for 3 months and Rosuvastatin (20mg daily) for at least 6 months as well as traditional risk factors management.
4. Patients were followed up for mRS score, stroke recurrence, medication compliance and laboratory examination including blood routine tests, liver functions and creatine kinase et al at 3 months, 6 months and 12 months after stroke onset. Additionally, patients are required to retake new HRMRI imaging of brain at 6 months.Remote patient education by We-Chat will be performed.
5. Our study aims to explore the stroke mechanisms of symptomatic intracranial atherosclerosis, the dynamic changes under aggressive medical treatment and their associations with clinical events using conventional MRI sequences plus HR-MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-80 years old
2. First-ever stroke patients confirmed by diffusion weighted imaging (DWI) attributed to intracranial artery stenosis (> 50%) within 7 days after onset.
3. Patients with stable vital signs.
4. Patients who have underwent thrombolytic/intravascular therapy are allowed to enroll in the study.

Exclusion Criteria:

1. Patients with > 50% ipsilateral carotid artery stenosis, cardiac embolism ,and any other stroke etiologies such as vasculitis, dissection or other causes.
2. Patients with absolute/relative contraindication to MRI (including but not confined to metal in the body and claustrophobia).
3. Patients who cannot comply with MRI exam.
4. Patients who decline the consent.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital based population
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
poor functional outcome | 90 day after stroke onset
  The Rankin Score runs from 0-6, running from perfect health without symptoms to death. mRS 0-2 are defined as favorable outcomes while mRS 3-6 as unfavorable outcomes.0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead.
Number of Participants with stroke recurrence | 12 months after stroke onset
  stroke recurrence with new lesions on DWI
Evolution of intracranial atherosclerosis burden | 6 months after stroke onset
  Changes of plaque and thrombus volume on HR-MRI images at the admission and the follow-up

SECONDARY OUTCOMES:
Number of Participants with Death due to Heart Disease, Cerebravascular Disease or Other Vascular Etiology | 12 months after stroke onset
  death due to stroke, intracranial hemorrhage,heart attack,heart failure, arrhythmia,pulmonary embolism,visceral hemorrhage or other vascular etiology

OTHER OUTCOMES:
Number of Participants with Adverse Events That Are Related to Anti-platelet Treatment | 12 months after stroke onset
  intracranial bleeding confirmed by CT，fatal bleeding causing hemodynamic abnormalities needed blood tranfusion or surgical intervention
Number of Participants with Adverse Events That Are Related to StatinTreatment | 12 months after stroke onset
  more than 3-fold liver enzyme increase，rhabdomyolysis

CONTACTS AND LOCATIONS:
Overall Officials: Weihai Xu, MD, Study Chair — Peking Union Medical College Hospital
Locations (38):
- China (38):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chao-Yang hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - General Hospital of Chinese Armed Police Forces, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - The first affiliated hospital affiliated to AMU (Southwest Hospital), Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The University of HongKong-Shenzhen Hospital, Shenzhen, Guangdong
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - Hong Xinglong Central Hospital, Shuangyashan, Heilongjiang
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - Affiliated Taihe Hospital of Hubei University of Medicine, Shiyan, Hubei
  - Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Subei People's Hospital of Jiangsu Province, Yangzhou, Jiangsu
  - China-Japan Union Hospital, Jilin University, Changchun, Jilin
  - General Hospital of Shen Yang Millitary Command, Shenyang, Liaoning
  - People's Hospital Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Shandong Provincial Hospital, Jinan, Shandong
  - JiNing NO.1 People Hospital, Jining, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Qilu Hospital of Shandong University (Qingdao), Qingdao, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Shanghai Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tongren Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Taiyuan Central Hospital of Shanxi Meidical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial Tongde Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Background] Li ML, Xu WH, Song L, Feng F, You H, Ni J, Gao S, Cui LY, Jin ZY. Atherosclerosis of middle cerebral artery: evaluation with high-resolution MR imaging at 3T. Atherosclerosis. 2009 Jun;204(2):447-52. doi: 10.1016/j.atherosclerosis.2008.10.019. Epub 2008 Oct 25. PMID 19041971
- [Background] Mazighi M, Labreuche J, Gongora-Rivera F, Duyckaerts C, Hauw JJ, Amarenco P. Autopsy prevalence of intracranial atherosclerosis in patients with fatal stroke. Stroke. 2008 Apr;39(4):1142-7. doi: 10.1161/STROKEAHA.107.496513. Epub 2008 Feb 28. PMID 18309170
- [Background] Xu WH, Li ML, Gao S, Ni J, Zhou LX, Yao M, Peng B, Feng F, Jin ZY, Cui LY. In vivo high-resolution MR imaging of symptomatic and asymptomatic middle cerebral artery atherosclerotic stenosis. Atherosclerosis. 2010 Oct;212(2):507-11. doi: 10.1016/j.atherosclerosis.2010.06.035. Epub 2010 Jun 25. PMID 20638663
- [Background] Xu WH, Li ML, Gao S, Ni J, Zhou LX, Yao M, Peng B, Feng F, Jin ZY, Cui LY. Plaque distribution of stenotic middle cerebral artery and its clinical relevance. Stroke. 2011 Oct;42(10):2957-9. doi: 10.1161/STROKEAHA.111.618132. Epub 2011 Jul 28. PMID 21799160
- [Background] Xu WH, Li ML, Gao S, Ni J, Yao M, Zhou LX, Peng B, Feng F, Jin ZY, Cui LY. Middle cerebral artery intraplaque hemorrhage: prevalence and clinical relevance. Ann Neurol. 2012 Feb;71(2):195-8. doi: 10.1002/ana.22626. PMID 22367991
- [Background] Xu WH, Li ML, Niu JW, Feng F, Jin ZY, Gao S. Intracranial artery atherosclerosis and lumen dilation in cerebral small-vessel diseases: a high-resolution MRI Study. CNS Neurosci Ther. 2014 Apr;20(4):364-7. doi: 10.1111/cns.12224. Epub 2014 Jan 15. PMID 24423003
- [Background] Xu WH, Li ML, Niu JW, Feng F, Jin ZY, Gao S. Deep tiny flow voids along middle cerebral artery atherosclerotic occlusions: a high-resolution MR imaging study. J Neurol Sci. 2014 Apr 15;339(1-2):130-3. doi: 10.1016/j.jns.2014.01.042. Epub 2014 Feb 6. PMID 24530171
- [Background] Li M, Wu SW, Xu WH. High-resolution MRI of radiation-induced intracranial vasculopathy. Neurology. 2015 Feb 10;84(6):631. doi: 10.1212/WNL.0000000000001223. No abstract available. PMID 25666631
- [Background] Derdeyn CP, Chimowitz MI, Lynn MJ, Fiorella D, Turan TN, Janis LS, Montgomery J, Nizam A, Lane BF, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Lynch JR, Zaidat OO, Rumboldt Z, Cloft HJ; Stenting and Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis Trial Investigators. Aggressive medical treatment with or without stenting in high-risk patients with intracranial artery stenosis (SAMMPRIS): the final results of a randomised trial. Lancet. 2014 Jan 25;383(9914):333-41. doi: 10.1016/S0140-6736(13)62038-3. Epub 2013 Oct 26. PMID 24168957
- [Background] Xu YY, Li ML, Gao S, Hou B, Sun ZY, Zhou HL, Feng F, Xu WH. Non-moyamoya vessel network formation along steno-occlusive middle cerebral artery. Neurology. 2016 May 24;86(21):1957-63. doi: 10.1212/WNL.0000000000002698. Epub 2016 Apr 27. PMID 27164677